CLINICAL TRIAL: NCT04097795
Title: Incremental Cost-utility Study on Prehabilitation for Colon Cancer Surgery in Older Patients
Brief Title: Incremental Cost-Utility Study on Prehabilitation Among Older Patients With Colorectal Cancer Undergoing Surgery
Acronym: PreColo CU
Status: Terminated | Type: Observational
Why Stopped: Inclusions lagged far behind
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leading the Change: Collaboration of health Insurers in the Netherlands (Unknown)
Responsible Party: Sponsor
Other Study IDs: PreColo CU
Record Dates: First submitted 2019-09-12; First posted 2019-09-20 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehabilitation: Patients aged 70 years and above or with an American Society of Anesthesiologists (ASA) score of III, who are scheduled for colorectal cancer surgery in one of the participating hospitals which offer prehabilitation.
  Interventions: Other: Prehabilitation
- No prehabilitation: Patients aged 70 years and above or with an American Society of Anesthesiologists (ASA) score of III, who are scheduled for colorectal cancer surgery in one of the participating hospitals which do not offer prehabilitation.

INTERVENTIONS:
Other: Prehabilitation — According to our definition, prehabilitation consists of exercise therapy during at least 2 weeks. This is combined with optimalisation of the patients' nutritional status at least 2 weeks before surgery.
  Groups: Prehabilitation

SUMMARY:
A prospective multicenter observational cost-utility study following older or high-risk patients with colorectal cancer with and without prehabilitation before surgery.

DETAILED DESCRIPTION:
This study will answer the question whether prehabilitation is cost-effective in colorectal cancer surgery among individual patients aged 70 years and above or patients with an American Society of Anesthesiologists (ASA) score of III. We also aim to identify factors facilitating or impairing implementation of prehabilitation such that it is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years or American Society of Anesthesiologists (ASA) score of III
* Scheduled for colorectal cancer surgery

Exclusion Criteria:

* Metastatic disease known preoperatively
* ASA IV score or higher
* Paralytic or immobilized patients (not capable to perform exercise)
* Prior use of neoadjuvant therapy for the same indication
* Not able or willing to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 70 years and above or patients with an ASA III score who are diagnosed with colorectal cancer and are scheduled for surgery as primary intervention will be recruited in the outpatient clinic of the surgery department of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L | 0-6 months
  Quality of life according to the EuroQol-5 dimensions-5 levels questionnaire. The 5 dimensions cover mobility, selfcare, daily activities, pain/discomfort and anxiety. All dimensions are rated on a 5 level scale ranging from 'I have no problems with ....(dimension)' to 'I am not able to/I am extremely...(dimension)'. The first option is considered 'better' and the latter as 'worse'.
Costs | 0-6 months
  From a societal perspective including health care consumption costs, patient out-of-pocket costs, and productivity losses of informal caregivers

SECONDARY OUTCOMES:
Number of deceased patients | 0-6 months
  Data on mortality will be assessed based on medical records.
Morbidity | 0-6 months
  Number and severity of complications will be assed based on medical records.
(I)ADL dependence by GARS | 0-6 months
  Dependence regarding (instrumental) acitivities of daily living ((I)ADL)according to the Gait Assessment Rating Scale (GARS). Several items with regard to self-reliance are scored according to the phrase 'I can do ....(item) completely independently.......'. Possible answers are 'Without any effort', 'with some effort', 'With a lot of effort', and 'Only with help from others'. The first is considered better and the latter as worse.
(I)ADL dependence by TOPICS-SF | 0-6 months
  Dependence regarding (instrumental) acitivities of daily living according toThe Older Persons and Informal Caregivers Survey Short form (TOPICS-SF) questionnaire for patients. This questionnaire contains GARS and EQ-5D amongst others and is spread throughout the questionnaire.
Return to normal activity | 0-6 months
  The return to normal activity (RNA) of patients is investigated by the different questionnaires listed above on several time-points. After surgery, we can examine the time within a time frame of 6 months that patients return to their normal activities.
Care-related burden among informal caregivers | 0-6 months
  The Older Persons and Informal Caregivers Survey Minimum Dataset (TOPICS-MDS) questionnaire for caregivers in which the domains 'self-reported health' (by RAND-36 health survey), 'quality of life' (by carerQol), 'hours of informal care' (number), and 'perceived burden' (on visual analog scale) are covered.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel G Olde Rikkert, MD PhD, Principal Investigator — Department of Geriatric Medicine, RadboudUmC
Locations (5):
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Radboudumc, Nijmegen
  - Streekziekenhuis Koningin Beatrix, Winterswijk

IPD SHARING:
Plan to Share IPD: Undecided